CLINICAL TRIAL: NCT01667848
Title: Warmed, Humidified Carbon Dioxide Insufflation vs Standard Carbon Dioxide in Laparoscopic Cholecystectomy: a Double-blinded Randomized Controlled Trial
Brief Title: Warmed, Humidified Carbon Dioxide Insufflation vs Standard Carbon Dioxide in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Klugsberger Bettina, Dr.med, Ludwig Boltzmann Institute for Operative Laparoscopy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCHE0909
Record Dates: First submitted 2012-07-27; First posted 2012-08-17 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Cholecystolithiasis
Keywords: pain
MeSH Terms: conditions — Cholecystolithiasis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group B: Insufflation with warm gas (Experimental): Insufflation with warmed, humidified carbon dioxide insufflation during laparoscopic cholecystectomy using the optitherm® device attached to the insufflation equipment in all of the patients but was only activated by the single scrub nurse in those patients randomized to group B.
  Interventions: Device: Optitherm® device activated
- group A: Insufflation with cold gas (Experimental): group A: Insufflation with cold gas during laparoscopic cholecystectomy, the use of Optitherm® device, which was attached to the insufflation equipment in all of the patients but was inactivated in group A
  Interventions: Device: Optitherm® device inactivated

INTERVENTIONS:
Device: Optitherm® device activated — The use of Optitherm® device, which was attached to the insufflation equipment in all of the patients but was only activated by the single scrub nurse in those patients randomized to group B.
  Other Names: Optitherm® device (Storz, Tuttlingen, Germany)
  Arms: group B: Insufflation with warm gas
Device: Optitherm® device inactivated — The use of Optitherm® device, which was attached to the insufflation equipment in all of the patients but was inactivated in group A.
  Other Names: Optitherm® device (Storz, Tuttlingen, Germany)
  Arms: group A: Insufflation with cold gas

SUMMARY:
The purpose of this study is to determine the effect of warmed, humidified carbon dioxide Insufflation vs standard carbon dioxide in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Patients undergoing warmed, humidified carbon dioxide (CO2) insufflation for laparoscopic cholecystectomy will have less postoperative pain than patients undergoing laparoscopic cholecystectomy with standard CO2 insufflation. The study design is a double-blind, prospective, randomized study comparing patients undergoing laparoscopic cholecystectomy with standard CO2 insufflation vs those receiving warmed, humidified CO2. Main variables included postoperative pain (rated with a visual analog scales) and analgesic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cholecystolithiasis

Exclusion Criteria:

* Clinical diagnosis of cholecystolithiasis with cholecystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Shamiyeh, Univ-Doz Dr, Study Chair — Ludwig Boltzmann Institute for Operative Laparoscopy, 2nd Surgical Department, Academic Teaching Hospital, AKH Linz
Locations (1):
- 2nd Surgical Department, Academic Teaching Hospital, AKH Linz, Linz, Upper Austria, Austria

REFERENCES:
- [Background] Farley DR, Greenlee SM, Larson DR, Harrington JR. Double-blind, prospective, randomized study of warmed, humidified carbon dioxide insufflation vs standard carbon dioxide for patients undergoing laparoscopic cholecystectomy. Arch Surg. 2004 Jul;139(7):739-43; discussion 743-4. doi: 10.1001/archsurg.139.7.739. PMID 15249406
- [Background] Sammour T, Kahokehr A, Hill AG. Meta-analysis of the effect of warm humidified insufflation on pain after laparoscopy. Br J Surg. 2008 Aug;95(8):950-6. doi: 10.1002/bjs.6304. PMID 18618870
- [Background] Yu TC, Hamill JK, Liley A, Hill AG. Warm, humidified carbon dioxide gas insufflation for laparoscopic appendicectomy in children: a double-blinded randomized controlled trial. Ann Surg. 2013 Jan;257(1):44-53. doi: 10.1097/SLA.0b013e31825f0721. PMID 22824858
- [Background] Nguyen NT, Furdui G, Fleming NW, Lee SJ, Goldman CD, Singh A, Wolfe BM. Effect of heated and humidified carbon dioxide gas on core temperature and postoperative pain: a randomized trial. Surg Endosc. 2002 Jul;16(7):1050-4. doi: 10.1007/s00464-001-8237-0. Epub 2002 Mar 26. PMID 12165821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approval from the local institutional ethics committee was obtained on June 2011. Between July 1st, 2011 and December 28nd, 2013, a total of 148 patients were scheduled for laparoscopic cholecystectomy at the General Hospital in Linz, Austria
Pre-assignment Details: Patients converted intraoperative to open cholecystectomy or those undergoing a concomitant procedure were excluded from the study. Irregularities of the study protocol (absence of rectal probe, missing consent form, conversion to open cholecystectomy) entailed in exclusion of the study. Patients with acute cholecystitis were excluded of the study.
Groups:
- Group A: Insufflation With Cold Gas: Insufflation with cold gas during laparoskopic cholecystectomy
- Group B: Insufflation With Warm Gas: Insufflation with warm gas during laparoscopic cholecystectomy
Period: Overall Study
Arm/Group | Group A: Insufflation With Cold Gas | Group B: Insufflation With Warm Gas
Started | 67 | 81
Completed | 67 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group B: Insufflation with warm gas during laparoskopic cholecystectomy
- Total: Total of all reporting groups
Arm/Group | Group A: Insufflation With Cold Gas | Group B | Total
Number analyzed (Participants) | 67 | 81 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.87 (14.44) | 55.68 (16.93) | 55.7 (15.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 57 | 103
  Male | 21 | 24 | 45
Region of Enrollment [Number; unit: participants]
  Austria | 67 | 81 | 148

OUTCOME MEASURES:

1. Primary Outcome: Pain (Rated With a Visual Analog Scale for Pain)
Description: postoperative pain (rated with a visual analog scale for pain) and analgesic requirements at operation day.
  The visual analog scale for pain ranged from 0-10 (0 is no pain, 10 is Maximum of pain)
Time Frame: operation day
Reporting Status: Not Posted

2. Secondary Outcome: Core Temperature
Time Frame: one day postoperativly
Reporting Status: Not Posted

3. Primary Outcome: Pain (Rated With a Visual Analog Scale for Pain)
Description: as for outcome 1
Time Frame: first postoperative day
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Group A: Insufflation With Cold Gas | Group B
Number analyzed (Participants) | 67 | 81
units on a scale 0-10 | 2.22 (0.97) | 1.92 (0.84)

4. Secondary Outcome: Core Temperature
Description: core temperature during laparoscopic cholecystectomy using a rectal probe
Time Frame: during operation
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Group A: Insufflation With Cold Gas | Group B
Number analyzed (Participants) | 67 | 81
degree celsius | 36.85 (0.46) | 37.07 (0.35)

ADVERSE EVENTS:
Groups:
- Group A: Insufflation with cold gas during laparoscopic cholecystectomy
- Group B: Insufflation with warm gas during laparoscopic cholecystectomy
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/81
Other Adverse Events (participants affected / at risk) | 0/67 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No